CLINICAL TRIAL: NCT06260774
Title: A Phase 1/2 Multicenter, Open-Label, Dose-escalation and Expansion Study of TTX-MC138 in Subjects With Advanced Solid Tumors
Brief Title: Study of TTX-MC138 in Subjects With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TransCode Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TTX-MC138-002; 1R44CA295173-01 (NIH)
Record Dates: First submitted 2023-12-12; First posted 2024-02-15 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Dose Escalation Study Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose level 1 (Experimental): 0.4 mg/kg of TTX-MC138
  Interventions: Drug: TTX-MC138
- Dose level 2 (Experimental): 0.8 mg/kg of TTX-MC138
  Interventions: Drug: TTX-MC138
- Dose level 3 (Experimental): 3.2 mg/kg of TTX-MC138
  Interventions: Drug: TTX-MC138

INTERVENTIONS:
Drug: TTX-MC138 — The starting dose of TTX-MC138 in the first cohort will be 0.4 mg/kg and will be increased incrementally in subsequent cohorts until maximum tolerated dose (MTD) determination.

SUMMARY:
A Phase 1/2 Multicenter, Open-Label, Dose-Escalation and Expansion Study of TTX MC138 in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
The study will consist of 2 phases, dose escalation and dose expansion, with 3 study periods: Screening (up to 28 days), Treatment (28-day treatment cycles, with dosing on Day 1), and Survival Follow-up (every 3 months). Each 28-day cycle is comprised of 1 dose of study drug administered as an intravenous (IV) infusion on Day 1.

A subject will continue on treatment until a dose limiting toxicity (DLT) is observed, other adverse event (AE) leading to unacceptable toxicity as assessed by the Investigator, progression of disease, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed diagnosis of relapsed/refractory metastatic or locally advanced solid tumor where no standard therapy exists, standard therapy has failed and have no available therapies with known clinical benefit.
2. Must have measurable or evaluable disease per RECIST version 1.1.
3. ≥18 years at the time of informed consent.
4. Life expectancy of ≥3 months
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2.
6. Have adequate organ function defined as:

   1. Platelet count ≥75×109/L with no platelet transfusions in the past 7 days
   2. Absolute neutrophil count ≥1.0×109/L
   3. Hemoglobin ≥8 g/dL (red blood cell transfusion may be used to reach 8 g/dL but must have been administered at least 1 week prior to the administration of the study drug)
   4. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <2.5× the upper limit of normal (ULN) if no hepatic metastases are present; <5× ULN if hepatic metastases are present
   5. Total bilirubin <1.5× ULN; <3 X ULN in the presence of Gilbert's disease
   6. Estimated (Cockcroft-Gault formula) or measured creatinine clearance ≥60 mL/min
   7. International normalized ratio (INR) ≤1.5× ULN unless participant is receiving anticoagulant therapy as long as the prothrombin time (PT) or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants
7. If female of childbearing potential, either abstain from sexual intercourse or employ highly effective contraception measures during the study and for ≥30 days after the administration of the study drug. Highly effective measures include 2 forms of contraception. Postmenopausal or surgically sterile women (ie, hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) are eligible. Postmenopausal status is defined as either: amenorrheic for ≥12 months following cessation of exogenous hormonal treatments and without an alternative medical cause; luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for women <50 years of age; radiation-induced ovarian ablation with last menses ≥1 year ago; or chemotherapy-induced menopause with a ≥1-year interval since last menses. Female subjects must refrain from donating or banking eggs (ova, oocytes) and retrieving eggs for use during study treatment and for 30 days after the administration of the study drug.
8. For male subjects not surgically sterile, must either abstain from sexual intercourse or employ highly effective contraception (condoms or other barrier forms of contraception) during the study and for at least 30 days after the administration of the study drug. Male subjects should also avoid semen donation or providing semen for in vitro fertilization during the above-mentioned duration.
9. Able to understand and willing to provide informed consent and able to comply with the study procedures, including biopsy, and restrictions.

Exclusion Criteria:

1. Unwilling or unable to comply with scheduled visits, study drug administration plan, laboratory tests, or other study procedures and study restrictions.
2. Have received anticancer therapy (including both systemic therapy and radiotherapy, but not including immunotherapy or other antibody therapies) within 14 days or 5 half-lives (whichever is shorter) of study drug administration or;

   a. received antibody therapy within 30 days before the start of study drug administration.
3. Have a history of a second primary malignancy that has been diagnosed or required active therapy within the past year.

   a. Note: The following prior malignancies are not exclusionary: completely resected basal cell and squamous cell skin cancer, curatively treated localized prostate or breast cancer, curatively treated localized thyroid cancer, and completely resected carcinoma in situ of any site.
4. Have central nervous system (CNS) metastases or primary CNS tumor that is associated with progressive neurologic symptoms or requires ongoing corticosteroids to control the CNS disease. Subjects must have a stable neurologic status without steroid support for ≥2 weeks before the start of study drug administration. Subjects with stable or asymptomatic CNS metastases or primary CNS are eligible.
5. Require treatment with traditional/herbal medicines or their preparations indicated for tumors or with adjuvant anti-tumor effects that cannot be discontinued during the study.
6. Have clinically significant, uncontrolled cardiovascular disease including congestive heart failure Class III or Class IV according to the New York Heart Association classification; myocardial infarction or unstable angina within the previous 6 months; uncontrolled hypertension (Grade ≥3); or clinically significant, uncontrolled arrhythmia, including bradyarrhythmia that may cause QT prolongation (eg, Type II second-degree heart block or third-degree heart block).
7. Have QT interval corrected using Fridericia's formula >480 msec. Unless the subject has a history of prolonged QT syndrome or torsade de pointes or a familial history of prolonged QT syndrome.
8. Have a history of acute ischemic stroke, diagnosed by imaging (CT or MRI) or clinical diagnosis within 6 months prior to screening.
9. Have any severe or uncontrolled systemic disease or condition per clinical judgement, including: (i) uncontrolled hypertension or diabetes; (ii) serious cardiac, pulmonary, or renal conditions; (iii) active bleeding diatheses; (iv) any active type of bacterial, viral, fungal, or other infection that would pose a significant risk to the subject in the opinion of the Investigator; (v) cerebrovascular accident within the last 6 months before administration of study drug.
10. Have received a major surgical procedure within 28 days before the start of study drug administration (procedures such as central venous catheter placement and tumor needle biopsy are not considered major surgical procedures). The study center should discuss other minor surgeries with the sponsor.
11. Clinical diagnosis of hemochromatosis or secondary iron overload,
12. Have known human immunodeficiency virus (HIV), hepatitis B virus, or hepatitis C virus infection that is not well-controlled and meets any of the following exclusion criteria:

    1. Documented detectable HIV RNA within 4 weeks of study drug administration,
    2. Acquired immunodeficiency syndrome defining opportunistic infections within the past 12 months prior to study enrollment, and
    3. Is not on antiretroviral therapy for at least 4 weeks prior to study enrollment.
13. Have clinical signs or symptoms consistent with COVID-19 infection or confirmed infection by appropriate laboratory test (done at the discretion of Investigator or per local regulation) within the last 2 weeks before the administration of the study drug. In case of confirmed COVID-19 infection before screening, documentation of resolution of infection by appropriate laboratory test is required.
14. Have received or are planning to receive a COVID-19 vaccination within 2 weeks before or after the administration of the study drug. However, COVID-19 vaccinations received >2 weeks before or after the administration of the study drug are permitted.
15. Have received a live or live attenuated vaccines within 30 days before the administration of the study drug.
16. Have any unresolved clinically relevant toxicities from prior therapy, greater than NCI CTCAE Grade 1 at the time of starting study treatment, except for alopecia.
17. Have a history of hypersensitivity to active or inactive excipients of the study drug or drugs with a similar chemical structure or class to the study drug, including ferumoxytol (Feraheme®).
18. Have an active autoimmune disease (eg, rheumatoid arthritis, systemic lupus erythematosus, ulcerative colitis, Crohn's disease, multiple sclerosis, ankylosing spondylitis, thyroiditis) requiring continuing immune suppressive therapy, including >10 mg prednisone per day or equivalent.
19. Pregnant or breastfeeding at the time of screening or on Day 1 before TTX-MC138 as documented by a serum beta human chorionic gonadotropin pregnancy test consistent with pregnancy.
20. Known current drug or alcohol abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation - Adverse Events | Throughout study treatment for 18 subjects, for average of 3 months and post treatment for survival follow-up through study completion, an average of 1 year
  The safety and tolerability of escalating dose levels of TTX-MC138 to determine incidence of treatment-emergent adverse events (TEAEs).
Dose Escalation - Overall Response Rate (ORR) | Throughout study treatment for 18 subjects, for average of 3 months and post treatment for survival follow-up through study completion, an average of 1 year
  proportion of subjects with a best response of CR, PR, or stable disease for at least 8 weeks per RECIST version 1.1.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mary Crowley Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - START Mountain Region, West Valley City, Utah
  - Next Oncology, Fairfax, Virginia